CLINICAL TRIAL: NCT04349462
Title: Post Critical Illness Dysphagia in the Intensive Care Unit (Dysphagia-ICU): a Single Centre Prospective Cohort Study
Brief Title: Post Critical Illness Dysphagia in the Intensive Care Unit
Acronym: DysphagiaICU
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment has been suspended during COVID19 Pandemic
Sponsor: St. Joseph's Healthcare Hamilton (Other)
Responsible Party: Principal Investigator, Waleed Al-Hazzani, Dr. Waleed Alhazzani, St. Joseph's Healthcare Hamilton
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 7298
Record Dates: First submitted 2020-04-14; First posted 2020-04-16 (Actual); Last update posted 2021-09-27 (Actual); Status verified 2021-09

CONDITIONS: Dysphagia
Keywords: Mehanical Ventilation, Dysphagia, VideoFluroscopy
MeSH Terms: conditions — Deglutition Disorders

STUDY DESIGN:
Intervention Model Description: Single center prospective pilot study of post critical illness dysphagia .
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- VFSS and Water Sip Test (Other): Enrolled patients will undergo a water sip test and Videofluroscopy Swallow Test (VFSS)
  Interventions: Diagnostic Test: VideoFlurosocopy Swallow Study; Diagnostic Test: Water Sip Test

INTERVENTIONS:
Diagnostic Test: VideoFlurosocopy Swallow Study — VFSS is a radiological examination that can identify the presence, nature and severity of any abnormalities in oropharyngeal, laryngeal and upper esophageal swallow physiology. The VFSS will be administered via a standardized protocol by a registered speech-language pathologist (SLP). During the VFSS, the patient is seated upright and swallows a variety of consistencies (eg. liquids, semisolids and solids) and volumes of barium-coated foods. A dynamic fluoroscopic image will be digitally captured and recorded.
  Other Names: VFSS
Diagnostic Test: Water Sip Test — The steps of the water sip test include; 1. The patient will be given 5 ml of water, and if tolerated 20 ml followed by 50 ml of water (thin fluid) and the patient is assessed for cough/chocking during or after swallowing, wet or weak cough after swallowing. 2. The patient is asked to produce sustained vowel /a/ before and after swallowing of water and voice change after swallowing will be observed and recorded.

SUMMARY:
The aims of the study are to determine: 1) the prevalence of ICU acquired dysphagia, 2) identify risk factors for ICU Acquired dysphagia, and 3) consequences of ICU acquired dysphagia including: ICU mortality, hospital mortality, days of mechanical ventilation, ICU length of stay, hospital length of stay, post extubation aspiration pneumonia, and rate of percutaneous endoscopic gastrostomy placed feeding tube (PEG-Tube) insertion, and/or total parenteral nutrition (TPN) and/or Dobhoff feeds.

DETAILED DESCRIPTION:
The RC will collect daily data on the use of advance life support, need for mechanical ventilation and outcomes (mortality, duration of mechanical ventilation, ICU length of stay, hospital length of stay). Enrolled patients will undergo a water sip test in the ICU and a videofluroscopic swallowing study (VFSS) performed by a registered speech-language pathologist (SLP). A VFSS is a videotaped or digitized dynamic fluoroscopic image that focuses on the oral, pharyngeal, laryngeal and upper esophageal swallow physiology. Patients will then be followed as two cohorts 1) patients that have dysphagia (or abnormal test) based on the VFSS, and 2) patients who have normal VFSS. We will then prospectively follow these two groups of patients during hospital stay censored at 30 days.

ELIGIBILITY:
Inclusion Criteria:

1. Adults (18 years of age and older)
2. Received mechanically ventilated for > 24 hours
3. Have been extubated for >24 hours
4. Hemodynamically stable (i.e. not requiring active resuscitation or vasoactive agents)
5. Able to participate in VFSS - with n the first 7 days after successful extubation. (+/- 2 days)

Exclusion Criteria:

1. Gastrostomy tube or a Gastro-jejunostomy tubes
2. Current contraindication to oral feeding (eg. recent gastrointestinal surgeries as indicated by their surgeons)
3. Being actively palliated
4. Tracheostomy
5. Neuromuscular condition associated with dysphagia: (e.g., amyotrophic lateral sclerosis, myasthenia gravis)
6. Pre-existing history of dysphagia
7. Ongoing respiratory support (defined as requiring ≥ 50% oxygen, bi-level positive airway pressure, or high flow nasal cannula) for 7 days or more after extubation.
8. Caring physician declined

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2019-09-04 (Actual); Primary Completion 2022-09 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Dysphagia | Hospital Discharge or 30 days post VFSS
  Defined as -abnormal VFSS scores resulting in need for modification of oral diet textures or non-oral means of nutrition and hydration provision.

SECONDARY OUTCOMES:
Aspiration | Hospital Discharge or 30 days post VFSS
  During drinking, eating, taking oral medication or other health professional-as documented in the clinical note by the treating physician
Pneumonia | Hospital Discharge or 30 days post VFSS
  Define as new pneumonia after extubation as noted in clinical chart
Length of Stay | Hospital Discharge or 30 days post VFSS
  ICU and Hospital
PEG tube insertion or need for TPF or Dobhoff feeds | Hospital Discharge or 30 days post VFSS
  • Percutaneous endoscopic gastrostomy placed feeding tube (PEG-Tube) insertion or need for TPF or Dobhoff feeds
Mortality | Hospital Discharge or 30 days post VFSS
  In ICU or In Hospital
Reintubation | Hospital Discharge or 30 days post VFSS
  Defined as reintubation within 30 days of original extubation during initial hospital admission. Reasons for reintubation will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Waleed Alhazzani, MD, MSc, Principal Investigator — McMaster University
Locations (1):
- St. Joseph's Healthcare Hamilton, Hamilton, Ontario, Canada